CLINICAL TRIAL: NCT06360861
Title: An Open-label, Non-randomized, Phase I Study of Allogeneic Placenta Derived Mesenchymal Stem Cells in Patients With Secondary-Progressive Multiple Sclerosis (SPMS),
Brief Title: Evaluate the Safety and Feasibility of Allogeneic Mesenchymal Stem Cells in Patients With Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1400-1-233-51589; IR.TUMS.MEDICINE.REC.1400.197 (Other Grant/Funding Number: Tehran University of Medical Sciences)
Record Dates: First submitted 2024-03-17; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis; Secondary-Progressive Multiple Sclerosis; Mesenchymal Stem Cells
Keywords: Mesenchymal Stem cells; Multiple Sclerosis; Placenta derived Mesenchymal Stem Cells; Stem Cell therapy; Neuroimmunology; Autoimmune Disease
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Open-label phase 1, single-center, pre-post comparison study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placenta derived mesenchymal cells (Experimental): Allogenic placenta derived mesenchymal stem cells, 3 million cells/kg body weight via intravenous injection
  Interventions: Biological: Allogenic placenta derived mesenchymal stem cells

INTERVENTIONS:
Biological: Allogenic placenta derived mesenchymal stem cells — Allogenic placenta derived mesenchymal stem cells, 3 million cells/kg body weight via intravenous injection.

SUMMARY:
To assess the safety and of a single dose of IV infusion of placenta derived Mesenchymal Stem Cells (PLMSCs) in patients with secondary progressive Multiple Sclerosis (SPMS) disease.

Monitoring will be encompassed baseline assessments and follow-ups over subsequent months, evaluating clinical signs, Expanded Disability Status Scale (EDSS), cytokines, diffusion tensor imaging (DTI), functional MRI (fMRI), cognitive & psychological evaluations, and flow cytometry for B cell markers.

DETAILED DESCRIPTION:
This open-label phase I study will be conducted in MS Clinic of Sina and Shariati Hospital of Tehran province .

In this study, diagnosis and management of MS patients will be performed based on McDonald's criteria and Iran's diagnostic and treatment protocols.

The patients will be received a single injection of PLMSCs through the intravenous cannula.

The proposed study will assess safety and short efficacy endpoints of PLMSCs administered to 5 patients with SPMS.

The primary objective of the trial is freedom from treatment associated adverse events at 1,3 and 6 months' post treatment. Secondary objective will be efficacy as assessed at baseline, at 1,3 and 6 months and will be based on the following: EDSS, cytokines, DTI, fMRI, cognitive & psychological evaluations, and flow cytometry for B cell markers.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Age between 17-45 years Patients with SPMS .
* Must be able to Sign informed consent .
* Currently taking Rituximab.
* Disease duration of more than 2 and less than 16 years.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* hepatitis B and C, human immunodeficiency virus (HIV), and human T-cell lymphotropic virus (HTLV) disease.
* Using cytotoxic agents within 3 months prior to the study.
* Severe anemia (hemoglobin< 8 mg/dl), coagulation disorders.
* history of malignancy .
* liver disorders .
* significant cardiac, renal or hepatic failure .
* Active or chronic infection.
* Life-threatening organ dysfunction.
* Unable to give written informed consent .
* Current treatment with an investigational therapy.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events [Safety and Tolerability]. | Up to 6 months
  adverse events

SECONDARY OUTCOMES:
Number of participants with a change in disability as measured by Expanded Disability Status Scale . | Up to 6 months
  Proportion of patients with clinical improvement in EDSS score compared to baseline. EDSS scores range from 0 = no disability to 10 = death due to MS and higher scores mean a worse outcome.
Number of participants with a change in cognitive function as measured by the Paced Auditory Serial Addition Test . | Up to 6 months
  The minimum score is 0 and maximum score is 60, and higher scores mean a better outcome.
Number of participants with a change in cognitive performance as measured by Persian version of minimal assessment of cognitive function in MS battery. | Up to 6 months
  Assessment of cognitive function
Number of participants with a change in brain connectivity as measured by Functional magnetic resonance imaging . | Up to 6 months
  Assessment of brain connectivity
Number of participants with a change in white matter integrity as measured by quantitative diffusion tensor imaging . | Up to 6 months
  Change from baseline in white matter integrity
Number of participants with a change in processing and motor speed as assessed by the Symbol Digit Modalities Test . | Up to 6 months
  Change from baseline in processing and motor speed of patients and higher scores mean a better outcome.
Number of participants with evaluation of verbal learning and memory deficits as measured by the California Verbal Learning Test second edition . | Up to 6 months
  Change from baseline in verbal learning and memory deficits and higher scores mean a better outcome.
Proportion of patients with change in CD20 / CD19 B cells surface markers | Up to 3 months
  Blood samples will be collected pre and post treatment for immediate or ulterior analysis.
Biological Assessments including IL-10, IL-6, IL-17, and TNFα levels of cytokines. | Up to 3 months
  Blood samples will be collected pre and post treatment for immediate or ulterior analysis.
Proportion of patients with change in T2 lesion volume on brain MRI. | Up to 6 months
  Change from baseline in T2 lesion volume.
Proportion of patients with change in brain volume on MRI. | Up to 6 months
  Change from baseline in brain volume
Proportion of patients for assessment of visuospatial learning as measured by the Brief Visuospatial Memory Test-Revised . | Up to 6 months
  Change from baseline in visuospatial learning
Proportion of patients for assessment of visuospatial ability as measured by Judgment of Line Orientation Test . | Up to 6 months
  Change from baseline in visuospatial ability
Proportion of patients for evaluation of executive functions as measured by the Delis-Kaplan Executive Function System Sorting and descriptive tests. | Up to 6 months
  Change from baseline in executive functions
Proportion of patients for measuring verbal fluency as measured by the Controlled Oral Word Association Test . | Up to 6 months
  Change from baseline in measuring verbal fluency
Proportion of patients for psychological assessment as measured by the validated Persian version of Symptom Checklist-90-Revised . | Up to 6 months
  Symptom Checklist-90(SCL-90) is a collection of nine subscales (with 90 items) for evaluation of Somatization, Obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism in the past week. Each item has a 5-point Likert scale and scoring from 0 to 4. SCL-90 Global Severity was calculated by dividing the sum of all subscales scores by 9.
Proportion of patients for evaluation of fatigue as measured by was examined by the Persian version of Fatigue Severity Scale . | Up to 6 months
  Fatigue Severity Scale(FSS )is a scale with 9 items, which assesses the fatigue severity in the past 2 weeks. Each item has a score from 1 to 7 and total score will be from 9 to 63. Higher FSS score indicates higher fatigue severity.
Proportion of patients for assessment of visuospatial ability as measured by the brief visuospatial memory test-revised test. | Up to 6 months
  Change from baseline in visuospatial ability
Proportion of patients for assessment of visuospatial ability as measured by the California Verbal Learning Test Second Edition test. | Up to 6 months
  Change from baseline in visuospatial ability

CONTACTS AND LOCATIONS:
Overall Officials: Abdorreza Naser Moghadasi, MD, Study Director — Multiple Sclerosis Research Center,Neuroscience Institute,Sina Hospital,Tehran, Iran.; Mohsen Nikbakht, PhD, Study Director — Research Institute for Oncology, Hematology& Cell Therapy Facility, Shariati Hospital ,Tehran, Iran.; Ameneh Shokati, PhD, Principal Investigator — Applied Cell Sciences,Tehran University of Medical Sciences,Tehran, Iran.
Locations (1):
- Tehran University of Medical Sciences,Tehran, Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shokati A, Naser Moghadasi A, Nikbakht M, Sahraian MA, Mousavi SA, Ai J. A focus on allogeneic mesenchymal stromal cells as a versatile therapeutic tool for treating multiple sclerosis. Stem Cell Res Ther. 2021 Jul 13;12(1):400. doi: 10.1186/s13287-021-02477-5. PMID 34256857
- [Background] Ebrahimi-Barough S, Ai J, Payab M, Alavi-Moghadam S, Shokati A, Aghayan HR, Larijani B, Arjmand B. Standard Operating Procedure for the Good Manufacturing Practice-Compliant Production of Human Endometrial Stem Cells for Multiple Sclerosis. Methods Mol Biol. 2021;2286:199-212. doi: 10.1007/7651_2020_281. PMID 32504294